CLINICAL TRIAL: NCT07022093
Title: Investigation of the Effects of Custom-Designed 3D-Printed and CAD-CAM-Produced Insoles in Individuals With Flexible Pes Planus
Brief Title: Effects of Custom-Designed 3D-Printed and CAD-CAM Insoles on Individuals With Flexible Flatfoot
Acronym: Insoles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GÖZDE KESİKBAŞ (Other Government)
Responsible Party: Sponsor-Investigator, GÖZDE KESİKBAŞ, Orthotic Prosthetist, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024211
Record Dates: First submitted 2025-05-31; First posted 2025-06-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pes Planus
Keywords: pes planus; 3D insoles; custom made insoles
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: Participants are allocated to two parallel groups for intervention and control, evaluated over the same study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom insoles manufactured using CNC technology (Active Comparator): Customised insoles will be produced using CNC technology and delivered based on the analyses of 20 patients with pes planus.
  Interventions: Device: Custom made insoles
- Custom insoles produced using 3D technology (Active Comparator): Custom insoles produced using 3D technology will be delivered to 20 patients with pes planus.
  Interventions: Device: Custom made insoles

INTERVENTIONS:
Device: Custom made insoles — For the production of insoles using the CAD-CAM method; In the production of insoles, medial longitudinal arch support will be added so that the subtalar joints are in a neutral position, and additionally, transverse arch support between 3.5-5 mm, lateral longitudinal arch support between 4-6 mm, and finger-under supports to assist with palmar grip will be designed in three dimensions using the EasyCad modelling interface. Using a Vulcan Computer Numerical Control (CNC) milling machine, the insoles will be machined from Ethylene Vinyl Acetate (EVA) material placed in blocks. After this process, the insoles will be adjusted on the milling machine to fit the patient's shoes.For the production of insoles using the 3D printing method, the Elegoo Neptune 4 Max 3D printer will be used. Using TPU material, medial longitudinal arch support will be added, along with transverse arch support between 3.5-5 mm, lateral longitudinal arch support between 4-6 mm, and finger support to aid palmar grip.
  Other Names: Insoles

SUMMARY:
This study aims to investigate the effects of custom-designed insoles produced using Computer Numerical Control (CNC) and 3D printers on plantar pressure distribution analysis, foot posture, plantar force distribution, foot pain, and satisfaction in patients diagnosed with pes planus.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the impact of custom-designed insoles, created using Computer Numerical Control (CNC) and 3D printing technologies, on plantar pressure distribution, foot posture, pain, and user satisfaction in individuals with flexible pes planus. The study targets adults aged 18-55, with specific clinical and postural inclusion criteria, and excludes individuals with biomechanical or neurological confounders.

Participants are randomly assigned to one of two intervention groups using a simple randomization method: one receiving CNC-produced insoles and the other 3D-printed insoles. Assessments are conducted before and after 8 weeks of insole use, employing standardized tools such as the Foot Posture Index, subtalar angle measurement, plantar pressure analysis, and satisfaction/function questionnaires. The primary aim is to explore comparative biomechanical and subjective outcomes to inform best practices in orthotic design and application.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 55 years
* Diagnosed with flexible pes planus (flat feet)
* No prior use of custom orthotic insoles within the past 6 months
* Able to walk independently without assistive devices
* Voluntarily agree to participate and provide informed consent

Exclusion Criteria:

* History of lower limb or foot surgery
* Presence of neurological, rheumatologic, or musculoskeletal disorders affecting gait
* Presence of severe foot deformities (e.g., rigid pes planus, cavus foot)
* Use of medications that affect muscle or joint function
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Change in Foot Function Index (FFI) Score | Baseline and 8 weeks after intervention
  This measure assesses changes in foot pain, disability, and activity limitation using the Foot Function Index (FFI). Participants complete the FFI questionnaire before and after the intervention period. The score ranges from 0 to 100, with higher scores indicating worse foot function.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Bek, PhD, Study Director — Lokman Hekim University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daryabor A, Kobayashi T, Saeedi H, Lyons SM, Maeda N, Naimi SS. Effect of 3D printed insoles for people with flatfeet: A systematic review. Assist Technol. 2023 Mar 4;35(2):169-179. doi: 10.1080/10400435.2022.2105438. Epub 2022 Aug 24. PMID 35882078
- [Background] Yarwindran, M., Sa'aban, N. A., Ibrahim, M., & Periyasamy, R. (2016). Thermoplastic elastomer infill pattern impact on mechanical properties 3D printed customized orthotic insole. ARPN J. Eng. Appl. Sci, 11(7).

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT07022093/Prot_SAP_ICF_000.pdf